CLINICAL TRIAL: NCT03467880
Title: Multicenter Study of Impulse Oscillometry in Chinese
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Collaborators: Beijing Hospital (Other Government); Beijing Children's Hospital (Other); Shanghai Zhongshan Hospital (Other); Second Affiliated Hospital, School of Medicine, Zhejiang University (Other); West China Hospital (Other); Tongji Hospital (Other); Third Military Medical University (Other); Xiangya Hospital of Central South University (Other); People's Hospital of Anshun City of Guizhou Province (Other); Shanghai Pulmonary Hospital, Shanghai, China (Other); Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Jinping Zheng, Vice-director, Guangzhou Institute of Respiratory Disease
Other Study IDs: GIRD201536
Record Dates: First submitted 2018-02-14; First posted 2018-03-16 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: Healthy Subjects; Chronic Obstructive Pulmonary Disease; Asthma; Interstitial Lung Disease; Upper Airway Obstruction
Keywords: Impulse Oscillometry; Chinese; Healthy Subjects; Chronic Obstructive Pulmonary Disease; Asthma; Interstitial Lung Disease; Upper Airway Obstruction; Reference Values
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Lung Diseases, Interstitial; Airway Obstruction | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (5):
- Healthy subjects: Healthy subjects.
  Interventions: Other: Clinical Observation
- Chronic obstructive pulmonary disease: Patience with chronic obstructive pulmonary disease.
  Interventions: Other: Clinical Observation
- Asthma: Patience with asthma.
  Interventions: Other: Clinical Observation
- Interstitial lung disease: Patience with interstitial lung disease.
  Interventions: Other: Clinical Observation
- Upper airway obstruction: Patience with upper airway obstruction.
  Interventions: Other: Clinical Observation

INTERVENTIONS:
Other: Clinical Observation — No treatment given but observation with IOS

SUMMARY:
The purpose of this study is to establish the reference values of impulse oscillometry (IOS) in healthy Chinese, and compare the indices of IOS in patients with lung disease, such as chronic obstructive pulmonary disease (COPD), asthma, interstitial lung disease (ILD), and upper airway Obstruction (UAO).

ELIGIBILITY:
Inclusion Criteria for healthy subjects:

* life-long non-smokers
* no symptoms and history of chronic cardiopulmonary diseases (chronic bronchitis, asthma, lung cancer, pulmonary fibrosis, pulmonary tuberculosis, chronic heart diseases, etc.)
* no abnormal findings on physical examination
* written informed consent was obtained

Inclusion Criteria for COPD:

* Diagnosis of chronic obstructive pulmonary disease (COPD), as classified by the Global Initiative for Chronic Obstructive Lung Disease (GOLD) guidelines and post-bronchodilator FEV1/FVC (forced vital capacity) < 70%.

Inclusion Criteria for asthma:

* Diagnosis of asthma, as classified by national and international asthma guidelines.

Inclusion Criteria for ILD:

* ILD diagnosis confirmed by lung biopsy, X ray or BALF analysis.

Inclusion Criteria for UAO:

* Diagnosis of UAO.

Exclusion Criteria for healthy subjects:

* upper or lower respiratory infection within 4 weeks
* long-term exposure to harmful gas or particles
* using β-blocker for treatment
* pregnant women, epileptic
* other diseases or surgeries potentially affecting lung function

Ages: 4 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be recruited from outpatient clinics.
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Airway resistance | one minute
  The indices of Airway resistance include total respiratory impedance (Zrs).

SECONDARY OUTCOMES:
forced vital capacity (FVC), forced expiratory volume in one second (FEV1), FEV1/FVC, and maximum midexpiratory flow (MMEF). | one minute
  The indices of spirometry include forced vital capacity (FVC), forced expiratory volume in one second (FEV1), FEV1/FVC, and maximum midexpiratory flow (MMEF).

CONTACTS AND LOCATIONS:
Overall Officials: Jinping Zheng, MD, Study Chair — State Key Laboratory of Respiratory Disease,China Clinical Research Center of Respiratory Disease, Guangzhou Institute of Respiratory Disease, First Affiliated Hospital of Guangzhou Medical University
Locations (2):
- China (2):
  - Beijing Hospital, Beijing
  - State Key Laboratory of Respiratory Disease,China Clinical Research Center of Respiratory Disease, Guangzhou Institute of Respiratory Disease, First Affiliated Hospital of Guangzhou Medical University, Guangzhou

REFERENCES:
- [Derived] Liang XL, Gao Y, Guan WJ, Du J, Chen L, Han W, Liu JM, Lu Y, Peng Y, Zhao BR, Wang T, Zheng JP. Reference values of respiratory impedance with impulse oscillometry in healthy Chinese adults. J Thorac Dis. 2021 Jun;13(6):3680-3691. doi: 10.21037/jtd-20-3376. PMID 34277060